CLINICAL TRIAL: NCT04526353
Title: Prospective Randomized Clinical Trial of Early Oxybutinin Treatment for Boys With Posterior Urethral Valves
Brief Title: Early Oxybutinin Treatment for Boys With Posterior Urethral Valves
Acronym: PRETIPUV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2018/65
Record Dates: First submitted 2020-07-29; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-07

CONDITIONS: Male Urogenital Diseases
Keywords: posterior urethral valves; urodynamic; anticholinergic
MeSH Terms: conditions — Male Urogenital Diseases | interventions — oxybutynin

STUDY DESIGN:
Intervention Model Description: Phase 2 non comparative randomized multicentre clinical trial with two parallel groups:
  * Oxybutynin (0.1 mg/kg twice daily) during 9 months.
  * No oxybutynin To determine whether the observed effects of oxybutynin are really due to the treatment we need to perform a randomized clinical trial. There is insufficient evidence in the literature about the natural evolution of the bladder in boys with PUV.
  Given the paucity of literature data, our objective is not to formally test the superiority of oxybutynin versus no drug but to detect and quantify the effect of oxybutynin. This is why our clinical is randomized but non-comparative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxybutynin during 9 months. (Experimental): 0.1mg / kg 2x / day from inclusion and for 9 months.
  Interventions: Drug: Oxybutynin 1 mg/ml Syrup
- No oxybutynin (No Intervention): No treatment affecting bladder function

INTERVENTIONS:
Drug: Oxybutynin 1 mg/ml Syrup — The Investigational Medicinal Product of this study is Oxybutynin 1 mg/ml Syrup (see Annex 1 for the Monograph of PMS-Oxybutynin provided by ANSM under the ATU.). It will be administered at the dose of 0.1 mg/kg/twice a day to patients randomized to the study treatment group. The dose will be adapted to the child's weight to the nearest kilogram.
  The recommended dosage for older children with neurologic bladder is 0.3 to 0.4mg/kg/day, whilst the dosage we will be using is effectively 0.2mg/kg/day. This is because we are taking into account the absence or pharmacological studies of oxybutynin use in children <1 year of age, as well as their specific liver metabolism. Furthermore, the dose of 0.1mg/kg twice daily is the dose used in children within the same age group in the study by Casey et al, 2012
  Arms: Oxybutynin during 9 months.

SUMMARY:
Boys with posterior urethral valves have bladder dysfunction of varying severity. Early treatment of these children with anticholinergics is recommended by some teams, although there have never been any clear studies on the subject. To our knowledge, no comparative study of the evolution of valve bladders with or without treatment has been carried out to date.

Anticholinergic treatment, although it may be beneficial in patients with abnormal bladder function, such as the neurologic bladders ( in Spina Bifida) for example, may have side effects and may not be of benefit for this valve population. The evolution of the valves could be spontaneously favorable.

This study would be the first randomized clinical trial of early therapeutic drug intervention in the posterior urethral valve population.

DETAILED DESCRIPTION:
Posterior urethral valves (VUPs) are the leading cause of subvesical obstruction in children with an incidence between 1 / 3,000 to 1 / 8,000 births. 25-45% of patients will have chronic renal failure and 10-20% will require a transplant. The association between long-term prognosis and bladder dysfunction is well known, leading many teams to suggest early initiation of treatment with anticholinergics.

However, this treatment has never been properly evaluated. In fact, a single study carried out in boys with valves taking oxybutynin from the age of 3 months to 2 years without a control group concluded that "the early use of anticholinergics in boys with VUP presenting high voiding pressures and low bladder capacity has a beneficial effect on bladder function. It is true that in children with neurologic bladders as in Spina Bifida, early treatment with anticholinergics seems to provide a benefit, but VUPs are not strictly speaking neurologic bladders. In addition, treatment with anticholinergics can have side effects and could even be harmful to the bladder, leading to myogenic bankruptcy. The only way to properly assess oxybutynin in this population is to conduct a prospective randomized study.

The proposed study includes a group treated with oxybutynin and a group without. Boys who have had valve resection for VUP within the first three months of life and who present an abnormal urodynamic assessment 3 months after valve resection will be included. Oxybutynin will be given at a dose of 0.1 mg / kg 2x / day, as syrup, in the treatment group. The control group will not have any treatment affecting bladder function. The pharmacokinetics of oxybutynin will be studied. Several urodynamic parameters including capacity or volume, voiding pressure and compliance will be studied. The objective is to perform a composite analysis that can reflect the complex functioning of the bladder. The children included will have urodynamics at the end of the study, after 9 months of treatment. The performance of urodynamic examinations will be standardized and there will be an external centralized analysis to validate the urodynamic results.

ELIGIBILITY:
Inclusion Criteria:

* Boys
* Aged 3 to 6 months
* Diagnosed with posterior urethral valves, and having undergone valve resection within the first 3 months of life
* Children who have had their valve resection at least 3 months before inclusion
* Having undergone urodynamic studies between 10 weeks and 6 months of age andshowing abnormal urodynamics, notably: high voiding pressure (>60cm H2O)/ small capacity bladder (<70% expected bladder volume)and for those without pop-off mechanisms, poor compliance (<10ml/cmH2O)/
* Holders of parental authority affiliated to French national health insurance
* With informed consent signed by holders of parental authority

Exclusion Criteria:

* Boys with posterior urethral valves and normal urodynamics or no urodynamic assessment
* Boys in whom urodynamic assessment is not possible for medical or anatomical reasons
* Boys requiring dialysis before the age of 3 months
* Contra-indication to oxybutynin such as hypersensitivity to oxybutynin or any of the excipients, digestive obstruction, occlusive or sub-occlusive syndrome, megacolon, digestive stasis, intestinal atony, paralytic ileus, ulcerative colitis, Hemorrhagic rectocolitis, Crohn's disease, Inflammatory bowel disease, Inflammatory organic colopathy, myasthenia, congenital glaucoma

Ages: 3 Months to 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Boys, aged 3 to 6 months, diagnosed with posterior urethral valves. Urethral valves (PUV) are the most common form of congenital urethral obstruction with an incidence ranging from 1/3,000 and 1/8,000 male births.
Enrollment: 50 (Estimated)
Dates: Start 2020-09-10 (Estimated); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
success of treatment defined by the association of the three events | 9 months after inclusion
  composite endpoints where the success of treatment at 9 months after inclusion is defined by the association of the three following events:
  * Voiding pressure <60 cmH2O AND
  * Bladder Volume ≥70% of theoretical value AND
  * for those without pop-off mechanisms, Bladder compliance >10mL/cmH2O A failure of treatment will be defined as the absence of at least one of these events.
  In presence of a pressure pop-off mechanism, only voiding pressure and bladder volume will be analyzed.

SECONDARY OUTCOMES:
Proportion of adverse events in each group | through study completion, an average of 9 months
Type of adverse events in each group | through study completion, an average of 9 months
  adverse event or serious adverse event
Incidence of urinary tract infections in each group | through study completion, an average of 9 months
Compliance with treatment | 9 months after inclusion
  Compliance with treatment will be evaluated through the proportion of oxybutynin treatment interruption
Sonographic changes | 9 months after inclusion
  Sonographic changes will be expressed as a degree of hydronephrosis at 12-15 months of life (9 months after inclusion)
Area under the plasma concentration versus time curve (AUC) of oxybutynin in treated boys over treatment | through study completion, an average of 9 months
  Area under the plasma concentration versus time curve (AUC) of oxybutinin in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Peak Plasma Concentration (Cmax) of oxybutynin in treated boys over treatment | through study completion, an average of 9 months
  Peak Plasma Concentration (Cmax) of oxybutynin in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Minimum plasma concentration (Cmin) of oxybutynin in treated boys over treatment | through study completion, an average of 9 months
  Minimum plasma concentration (Cmin) of oxybutynin in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Half-life of oxybutynin in treated boys over treatment | through study completion, an average of 9 months
  Half-life of oxybutynin in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Area under the plasma concentration versus time curve (AUC) of desethyloxybutynin (metabolite) in treated boys over treatment | through study completion, an average of 9 months
  Area under the plasma concentration versus time curve (AUC) of desethyloxybutynin (active metabolite) in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Peak Plasma Concentration (Cmax) of desethyloxybutynin (metabolite) in treated boys over treatment | through study completion, an average of 9 months
  Peak Plasma Concentration (Cmax) of desethyloxybutynin (active metabolite) in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Minimum plasma concentration (Cmin) of desethyloxybutynin (metabolite) in treated boys over treatment | through study completion, an average of 9 months
  Minimum plasma concentration (Cmin) of desethyloxybutynin (active metabolite) in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
Half-life of desethyloxybutynin (metabolite) in treated boys over treatment | through study completion, an average of 9 months
  Half-life of desethyloxybutynin (active metabolite) in treated boys over treatment. Pharmacokinetic samples (6 points from Cmin to H+3h) at 2 weeks, 3 and 9 months after inclusion will be used to study and determine the pharmacokinetic parameters. In order to avoid having to take blood sample from the child several times, it is proposed to use a small venous catheter during the time of the pharmacokinetic samples
creatinine clearance in each group | through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent L FOURCADE, MD, Principal Investigator — University Hospital, Limoges; Alice A FAURE, MD, Principal Investigator — APHM - Hôpital Timone Enfants; Thomas BLANC, MD, Principal Investigator — APHP - Hôpital Necker Enfants Malades; Alaa A EL GHONEIMI, MD, Principal Investigator — APHP- Hôpital Robert Debré; Alexis A ARNAUD, MD, Principal Investigator — Rennes University Hospital; Ourdia O BOUALI, MD, Principal Investigator — University Hospital, Toulouse; Jean-Baptiste JB MARRET, MD, Principal Investigator — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casey JT, Hagerty JA, Maizels M, Chaviano AH, Yerkes E, Lindgren BW, Kaplan WE, Meyer T, Cheng EY. Early administration of oxybutynin improves bladder function and clinical outcomes in newborns with posterior urethral valves. J Urol. 2012 Oct;188(4 Suppl):1516-20. doi: 10.1016/j.juro.2012.03.068. Epub 2012 Aug 19. PMID 22910256